CLINICAL TRIAL: NCT03237377
Title: Neoadjuvant Immunoradiation for Stage III Resectable Non-Small Cell Lung Cancer
Brief Title: Neoadjuvant Immunoradiation for Resectable Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J1772; IRB00127418 (Other: JHM IRB); ESR-16-12244 (Other: AstraZeneca)
Record Dates: First submitted 2017-07-19; First posted 2017-08-02 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; tremelimumab; Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Durvalumab with Radiation (Experimental): Drug: Durvalumab Other Names: MEDI4736
  MEDI4736 1500mg via IV infusion every 4 weeks for up to 3 doses/cycles Intervention: Radiation: Thoracic Radiation 5 days per week in once daily fractionation, 1.8-2.0 Gy per fraction
  Intervention: Procedure/Surgery: lobectomy patients may proceed to surgery post drug and radiation intervention for lung lobectomy
  Intervention: Drug: Standard of care adjuvant chemotherapy patients may or may not proceed to adjuvant chemotherapy post trial drug and radiation intervention and surgery
  Interventions: Drug: Durvalumab; Radiation: Thoracic Radiation; Procedure: lobectomy; Drug: Standard of care adjuvant chemotherapy
- Durvalumab and Trememlimumab with Radiation (Experimental): Drugs: Durvalumab + Tremelimumab Other Names: MEDI4736 and CP-675 MEDI4736 1500mg via IV infusion every 4 weeks for up to 3 doses/cycles + CP-675 206 75mg via IV infusion every 4 weeks up 3 doses/cycles Intervention: Radiation: Thoracic Radiation 5 days per week in once daily fractionation, 1.8-2.0 Gy per fraction Intervention: Procedure/Surgery: lobectomy patients may proceed to surgery post drug and radiation intervention for lung lobectomy
  Intervention: Drug: Standard of care adjuvant chemotherapy patients may or may not proceed to adjuvant chemotherapy post trial drug and radiation intervention and surgery
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Thoracic Radiation; Procedure: lobectomy; Drug: Standard of care adjuvant chemotherapy

INTERVENTIONS:
Drug: Durvalumab — 1500mg via IV infusion every 4 weeks for up to 3 doses/cycles
  Other Names: [MEDI4736]
Drug: Tremelimumab — 75mg via IV infusion every 4 weeks
  Other Names: [CP-675 206]
  Arms: Durvalumab and Trememlimumab with Radiation
Radiation: Thoracic Radiation — 5 days per week in once daily fractionation, 1.8-2.0 Gy per fraction
Procedure: lobectomy — patients may proceed to surgery post drug and radiation intervention for lung lobectomy
Drug: Standard of care adjuvant chemotherapy — patients may or may not proceed to adjuvant chemotherapy post trial drug and radiation intervention and surgery

SUMMARY:
This is a pilot study of neoadjuvant 'immunoradiation' (durvalumab or durvalumab plus tremelimumab) administered every 4 weeks for 2 doses, concurrently with standard thoracic radiation (RT) (45Gy in 25 fractions), with one dose of immunotherapy alone delivered in the pre-surgical window, prior to surgical resection, for patients with stage IIIA NSCLC that is deemed resectable with a lobectomy by a thoracic surgeon. If preliminary safety of the durvalumab/thoracic RT combination is established, a second cohort investigating the combination of durvalumab/tremelimumab/thoracic RT prior to surgical resection will be opened. After surgical resection, patients may receive standard adjuvant chemotherapy, as deemed appropriate by the treating investigator.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization obtained.
* Histologically-confirmed diagnosis of stage III non-small cell lung cancer (NSCLC)
* Age≥18 years
* Life expectancy >6 months
* Body weight >30kg
* Subjects with non-small cell lung cancer deemed surgically resectable by an attending thoracic surgeon with lobectomy
* ECOG Performance Status 0-1
* Normal bone marrow and organ function on routine laboratory tests, as defined in section 4.1
* Evidence of post-menopausal status or negative urinary/serum pregnancy test for female pre-menopausal subjects. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
* Ability to understand and willingness of sign consent form
* Willingness to comply with the protocol for the duration of the study

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (includes AstraZeneca staff and staff at the study site)
* Prior investigational therapy within 28 days/at least 5 half-lives before study drug administration
* Prior chest radiation
* Prior history of interstitial lung disease or pneumonitis requiring corticosteroids, or active non-infectious pneumonitis
* Patients only suitable for surgical management with pneumonectomy, deemed by an attending thoracic surgeon
* Prior therapy with PD-1, PD-L1, CTLA-4 or anti-cancer vaccines, including durvalumab and tremelimumab
* Participation in another clinical study with an investigational product in the last 4 weeks or equivalent of 5 half-lives of the first dose of study treatment, whichever is shorter
* History of another primary malignancy that requires active ongoing treatment or, in the opinion of the investigator, is likely to require treatment within 6 months of trial enrollment
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Any unresolved toxicity (>CTCAE grade 2) from previous anti-cancer therapy
* Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion (vitiligo or alopecia; hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement; any chronic skin condition that does not require systemic therapy; active disease in the last 5 years may be included but only after consultation with the study physician; celiac disease controlled by diet alone.)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study result.
* Known allergy or hypersensitivity to IP or any excipient
* Uncontrolled psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written consent
* Any condition that, in the opinion of the investigator would interfere with evaluation of study treatment or interpretation of patient safety or study results.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Forde, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated due to low accrual on Arm A (Durvalumab with Radiation) so no participants were assigned to Arm B (Durvalumab and Trememlimumab with Radiation).
Groups:
- Durvalumab With Radiation: Drug: Durvalumab Other Names: MEDI4736
  MEDI4736 1500mg via IV infusion every 4 weeks for up to 3 doses/cycles Intervention: Radiation: Thoracic Radiation 5 days per week in once daily fractionation, 1.8-2.0 Gy per fraction
  Intervention: Procedure/Surgery: lobectomy patients may proceed to surgery post drug and radiation intervention for lung lobectomy
  Intervention: Drug: Standard of care adjuvant chemotherapy patients may or may not proceed to adjuvant chemotherapy post trial drug and radiation intervention and surgery
  Durvalumab: 1500mg via IV infusion every 4 weeks for up to 3 doses/cycles
  Thoracic Radiation: 5 days per week in once daily fractionation, 1.8-2.0 Gy per fraction
  lobectomy: patients may proceed to surgery post drug and radiation intervention for lung lobectomy
  Standard of care adjuvant chemotherapy: patients may or may not proceed to adjuvant chemotherapy post trial drug and radiation intervention and surgery
- Durvalumab and Trememlimumab With Radiation: Drugs: Durvalumab + Tremelimumab Other Names: MEDI4736 and CP-675 MEDI4736 1500mg via IV infusion every 4 weeks for up to 3 doses/cycles + CP-675 206 75mg via IV infusion every 4 weeks up 3 doses/cycles Intervention: Radiation: Thoracic Radiation 5 days per week in once daily fractionation, 1.8-2.0 Gy per fraction Intervention: Procedure/Surgery: lobectomy patients may proceed to surgery post drug and radiation intervention for lung lobectomy
  Intervention: Drug: Standard of care adjuvant chemotherapy patients may or may not proceed to adjuvant chemotherapy post trial drug and radiation intervention and surgery
  Durvalumab: 1500mg via IV infusion every 4 weeks for up to 3 doses/cycles
  Tremelimumab: 75mg via IV infusion every 4 weeks
  Thoracic Radiation: 5 days per week in once daily fractionation, 1.8-2.0 Gy per fraction
  lobectomy: patients may proceed to surgery post drug and radiation intervention for lung lobectomy
  Standard of care adjuvant chemotherapy: patients may or may not proceed to adjuvant chemotherapy post trial drug and radiation intervention and surgery
Period: Overall Study
Arm/Group | Durvalumab With Radiation | Durvalumab and Trememlimumab With Radiation
Started | 9 | 0
Completed | 9 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The protocol planned for a second cohort for patients to be treated with durvalumab and trememlimumab with radiation, however, due to low accrual in cohort 1, there was no second cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab With Radiation | Durvalumab and Trememlimumab With Radiation | Total
Number analyzed (Participants) | 9 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 6 |  | 6
Age, Continuous [Mean (Full Range); unit: years] | 66 [45 to 77] |  | 66 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 |  | 5
  Male | 4 |  | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Non-Hispanic | 4 |  | 4
  Race/Ethnicity: White Ethnicity Unknown | 1 |  | 1
  Race/Ethnicity: Black/African-American Non-Hispanic | 1 |  | 1
  Race/Ethnicity: Asian Non-Hispanic | 1 |  | 1
  Race/Ethnicity: Race/Ethnicity Unknown | 2 |  | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 |  | 3
  United States | 6 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Toxicities as Measured by Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing adverse events as defined by CTCAE v4.0.
Time Frame: 3 months post surgery
Population: all participants who were assigned to the durvalumab with radiation arm
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab With Radiation | Durvalumab and Trememlimumab With Radiation
Number analyzed (Participants) | 9 | 0
Participants | 9 | 0

2. Primary Outcome: Feasibility of Preoperative Immunoradiation
Description: Number of participants with stage III resectable NSCLC who received durvalumab or durvalumab plus tremelimumab concurrently with thoracic radiation (RT) in the pre-surgical window prior to surgical resection, for whom planned surgical resection was not delayed.
Time Frame: Up to 3 years
Population: The study closed early due to low accrual on Arm A Durvalumab with Radiation so no data was collected for Arm B Durvalumab and Trememlimumab with Radiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab With Radiation | Durvalumab and Trememlimumab With Radiation
Number analyzed (Participants) | 9 | 0
Participants | 9 | 0

3. Secondary Outcome: Surgical Morbidity and Mortality
Description: Number of participants who experience post-operative death. Calculated through log-rank test and Cox proportional hazards (PH) model. The values in the table represent the number of participants who experienced post-operative death.
Time Frame: Up to 3 months post-surgery
Population: The study closed to enrollment before patients could be enrolled onto Arm B: durvalumab and trememlimumab with radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab With Radiation | Durvalumab and Trememlimumab With Radiation
Number analyzed (Participants) | 9 | 0
Participants | 0 | 0

4. Secondary Outcome: Percentage of Participants With Pathologic Response
Description: Percentage of participants with major pathologic response (MPR), partial response (PR) or no response (NR), where MPR is >90% reduction in tumor cells, PR = 10-90% or NR = 0-10%. The percentage of patients whose tumor samples achieve MPR, PR and NR will be tabulated.
Time Frame: Up to 3 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab With Radiation | Durvalumab and Trememlimumab With Radiation
Number analyzed (Participants) | 9 | 0
Participants | 9 | 0

5. Secondary Outcome: Percentage of Participants With Radiologic Response
Description: Percentage of participants with complete response (CR), partial response (PR), progressive disease (PD), and stable disease (SD) as defined by RECIST 1.1 and immune-related RECIST criteria when treated with preoperative immunoradiation followed by surgery. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, PD is >20% increase in sum of diameters of target lesions, SD is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: Up to 3 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab With Radiation | Durvalumab and Trememlimumab With Radiation
Number analyzed (Participants) | 9 | 0
Participants | 7 | 0

6. Secondary Outcome: Duration of Response as Measured by Recurrence-free Survival
Description: Time from first evidence of response until recurrence when treated with preoperative immunoradiation followed by surgery. Calculated through log-rank test and Cox proportional hazards (PH) model.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2026-01

7. Secondary Outcome: Overall Survival
Description: Number of months alive after treatment with preoperative immunoradiation followed by surgery. Calculated through log-rank test and Cox proportional hazards (PH) model.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: Post-surgery, up to 3 months.
Description: The number of participants at risk for SAEs, AEs, and all-cause mortality is zero for the Durvalumab and Trememlimumab With Radiation arm because the study was terminated and there were no patients enrolled onto arm B, and no data was collected.
Arm/Group | Durvalumab With Radiation | Durvalumab and Trememlimumab With Radiation
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/9 | 0/0
Other Adverse Events (participants affected / at risk) | 9/9 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab With Radiation (N=9) | Durvalumab and Trememlimumab With Radiation (N=0)
aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) — pulmonary embolism
appendicitis (Infections and infestations) | 1 (1) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab With Radiation (N=9) | Durvalumab and Trememlimumab With Radiation (N=0)
fatigue (General disorders) | 5 (5) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
facial pain (General disorders) | 1 (1) | 0 (0)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
thrombophelbitis (Vascular disorders) | 1 (1) | 0 (0)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)
fever (General disorders) | 1 (1) | 0 (0)
chills (General disorders) | 1 (2) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
violaceus raticular rash - upper forearm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
erythematous rash - thighs and knees (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
anterior chest rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sinus disorder - sinus drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
orange-colored skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pain at thoracotomy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (2) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 0 (0)
serum amylase increased (Investigations) | 1 (1) | 0 (0)
white blood cell decreased (Investigations) | 1 (1) | 0 (0)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT03237377/Prot_SAP_000.pdf